CLINICAL TRIAL: NCT04790370
Title: A Randomized Trial of Ultrasound-facilitated, Catheter-directed, Thrombolysis Versus Anticoagulation for Acute Intermediate-high Risk Pulmonary Embolism: The Higher-risk Pulmonary Embolism Thrombolysis Study
Brief Title: Ultrasound-facilitated, Catheter-directed, Thrombolysis in Intermediate-high Risk Pulmonary Embolism
Acronym: HI-PEITHO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: National PERT Consortium, Inc. (Unknown); University Medical Center Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2479
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
Keywords: Acute intermediate-high risk pulmonary embolism; Ultrasound-facilitated, catheter-directed thrombolysis; Thrombolysis
MeSH Terms: conditions — Pulmonary Embolism | interventions — Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Outcomes Assessor
Masking Description: Blinded adjudication of primary composite outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anticoagulation (Active Comparator): Low-molecular weight heparin (LMWH) or unfractionated heparin (UFH)
  Interventions: Drug: Anticoagulation with heparin
- Anticoagulation and EkoSonicTM Endovascular System (Active Comparator): Low-molecular weight heparin (LMWH) or unfractionated heparin (UFH) and EkoSonicTM Endovascular System [ultrasound-facilitated catheter-directed delivery of thrombolytic: 2 mg bolus/catheter + 1 mg/hour/catheter for 7 hours (total of 9 or 18 mg]
  Interventions: Drug: Anticoagulation with heparin; Device: EkoSonicTM Endovascular System

INTERVENTIONS:
Drug: Anticoagulation with heparin — Low-molecular weight heparin (LMWH) or unfractionated heparin (UFH)
  Other Names: heparin, LMWH, UFH, anticoag, antiplatelet
Device: EkoSonicTM Endovascular System — EkoSonicTM Endovascular System [ultrasound-facilitated catheter-directed delivery of thrombolytic: 2 mg bolus/catheter + 1 mg/hour/catheter for 7 hours (total of 9 or 18 mg]
  Other Names: EKOS, USCDT, CDT, thrombolysis, fibrinolysis
  Arms: Anticoagulation and EkoSonicTM Endovascular System

SUMMARY:
There are many available treatments for pulmonary embolism (PE), but the best treatment for this condition is not known. The HI-PEITHO study will compare two treatment options that are both available on the market for the treatment of PE.

Patients will be randomized 1:1 to receive either blood thinners (anticoagulation) or blood thinners (anticoagulation) in combination with a device called the EkoSonicTM Endovascular device to dissolve blood clots. Patients will be followed for 12 months after randomization and have assessments while in the hospital as well as at 7 days, 30 days, 6 months and 12 months after randomization. The study will try to find out if one of these treatments is better than the other at reducing the risk of death and other serious problems.

DETAILED DESCRIPTION:
This study will assess whether ultrasound-facilitated, catheter-directed thrombolysis and standard anticoagulation are associated with a significant reduction in the composite outcome of pulmonary embolism (PE)-related mortality, cardiorespiratory decompensation or collapse, or nonfatal symptomatic and objectively confirmed recurrence of PE compared to anticoagulation alone within seven days of randomization

The HI-PEITHO study has been designed to address the important gaps in clinical evidence by comparing the clinical benefit of the ultrasound-facilitated local delivery of a low dose thrombolytic agent and anticoagulation with those of anticoagulation alone in patients with intermediate-high risk PE at a higher estimated risk of early decompensation based on clinical parameters at presentation.

This study has a focus on improving the safety of thrombolysis and advancing the concept of intermediate-high risk and the PE severity criteria, to better identify patients who may clinically benefit from thrombolysis.

The results of this study will contribute further evidence to the existing data on the treatment and outcomes of acute, intermediate-high risk PE and provide controlled data related to catheter-based interventions.

Data will be entered by the site into an electronic database. The database will include data checks to compare data entered into the database against predefined rules for ranges and consistency with other data fields in the database.

Site monitoring will take place with source data verification to assess the accuracy and completeness of registry data by comparing the data to medical records and study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, inclusive
* Objectively confirmed acute PE, based on computed tomography pulmonary angiography (CTPA) showing a filling defect in at least one main or proximal lobar pulmonary artery
* Elevated risk of early death/hemodynamic collapse, indicated by at least two of the following new-onset clinical criteria:

  1. ECG-documented tachycardia with heart rate ≥100 beats per minute, not due to hypovolemia, arrhythmia, or sepsis;
  2. SBP ≤ 110 mm Hg for at least 15 minutes;
  3. respiratory rate > 20 x min^-1 or oxygen saturation on pulse oximetry (SpO2) < 90% (or partial arterial oxygen pressure < 60 mmHg) at rest while breathing room air;
* Right-to-left ventricular (RV/LV) diameter ratio ≥ 1.0 on CTPA
* Serum troponin I or T levels above the upper limit of normal
* Signed informed consent

Exclusion Criteria:

* Hemodynamic instability*, i.e. at least one of the following present:

  1. cardiac arrest or need for cardiopulmonary resuscitation;
  2. need for ECMO, or ECMO initiated before randomization
  3. PE-related shock, defined as: (i) SBP < 90 mmHg, or vasopressors required to achieve SBP ≥ 90 mmHg, despite an adequate volume status; and (ii) end-organ hypoperfusion (altered mental status; oliguria/anuria; increased serum lactate);
  4. isolated persistent hypotension (SBP < 90 mmHg, or a systolic pressure drop by at least 40 mmHg for at least 15 minutes), not caused by new-onset arrhythmia, hypovolemia, or sepsis * Patients who presented with temporary need for fluid resuscitation and/or low-dose catecholamines may be included, provided that they could be stabilized within 2 hours of admission and maintain SBP of ≥ 90 mmHg and adequate organ perfusion without catecholamine infusion.
* Need for admission to an intensive care unit for a reason other than the index PE episode. NB: Patients who test positive for SARS-CoV-2 can be enrolled where the investigator believes that the pulmonary embolism is the dominant pathology in the patient's clinical presentation and qualifying cardiorespiratory parameters.
* Temperature above 39 degrees C / 102.2 degrees F
* Logistical reasons limiting the rapid availability of interventional procedures to treat acute PE (e.g., during the outbreak of an epidemic)
* Index PE symptom duration > 14 days
* Active bleeding
* History of intracranial or intraocular bleeding at any time
* Stroke or transient ischemic attack within the past 6 months, or previous stroke at any time if associated with permanent disability
* Central nervous system neoplasm, or metastatic cancer
* Major neurologic, ophthalmologic, abdominal, cardiac, thoracic, vascular or orthopedic surgery or trauma (including syncope-associated with head strike or skeletal fracture) within the past 3 weeks
* Platelet count < 100 x 10^9 x L^-1
* Patients who have received a once-daily therapeutic dose of LMWH or a therapeutic dose of fondaparinux within 24 hours prior to randomization
* Patients who have received one of the direct oral anticoagulants apixaban or rivaroxaban within 12 hours prior to randomization
* Patients who have received one of the direct oral anticoagulants dabigatran or edoxaban for the index PE episode, as these drugs are not approved for patients who have not received heparin for at least 5 days
* Administration of a thrombolytic agent or a glycoprotein IIb/IIIa receptor antagonist during the current hospital stay and/or within 30 days, for any reason
* Chronic treatment with antiplatelet agents other than low-dose acetylsalicylic acid or clopidogrel 75 mg once daily (but not both). Dual antiplatelet therapy is excluded.
* Chronic treatment with a direct oral anticoagulant (apixaban, dabigatran, edoxaban or rivaroxaban)
* Chronic treatment with a vitamin K antagonist, or known coagulopathy including severe hepatic dysfunction, with an International Normalized Ratio (INR) > 1.5
* Pregnancy or lactation
* Previous inclusion in the study
* Known hypersensitivity to alteplase, LMWH or UFH, or to any of the excipients
* Life expectancy less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
PE-related mortality | Within seven days of randomization
  death resulting from PE
PE recurrence | Within seven days of randomization
  nonfatal symptomatic and objectively confirmed recurrence of PE
Cardiorespiratory decompensation or collapse | Within seven days of randomization
  Cardiorespiratory collapse or decompensation is defined as at least one of the following criteria:
  1. cardiac arrest or need for CPR at any time between randomization and day 7;
  2. signs of shock: new-onset persistent arterial hypotension (systolic blood pressure (SBP) below 90 mmHg or SBP drop by at least 40 mm Hg, over at least 15 minutes and despite an adequate volume status; or need for vasopressors to maintain SBP of at least 90 mmHg), accompanied by end-organ hypoperfusion (altered mental status; oliguria/anuria; or increased serum lactate) at any time between randomization and day 7;
  3. placement on extracorporeal membrane oxygenation (ECMO) at any time between randomization and day 7;
  4. intubation, or initiation of noninvasive mechanical ventilation at any time between randomization and day 7;
  5. National Early Warning Score (NEWS) of 9 or higher, between 24 hours and 7 days after randomization, confirmed on consecutive measurements taken twice, 15 minutes apart.

OTHER OUTCOMES:
Change in the RV-to-LV diameter ratio as measured by echocardiography | Between baseline and 48±6 hours
PE-related death | Within 7 days
  Death cause by pulmonary embolism (PE)
Cardiorespiratory decompensation | Within 7 days
Placement on ECMO or mechanical ventilation | Within 7 days
GUSTO major (moderate and severe) bleeding | Within 7 days
  Major bleeding will be adjudicated according to the GUSTO criteria:
  1. GUSTO severe or life-threatening bleeding: A bleeding episode that leads to hemodynamic compromise requiring emergency intervention (such as replacement of fluid and/or blood products, inotropic support, or surgical treatment), or is life-threatening or fatal.
  2. GUSTO moderate bleeding (a bleeding episode requiring blood transfusion(s), but which is not deemed life-threatening and does not lead to hemodynamic compromise requiring emergency fluid replacement, inotropic support, or interventional treatment) .
International Society on Thrombosis and Hemostasis (ISTH) major bleeding | Within 7 days, 30 days, and 6 months
  Major bleeding will also be adjudicated according to the ISTH criteria:
  1. Fatal bleeding and/or
  2. Symptomatic bleeding in a critical area or organ (intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome) and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (2 g/dL) or more, or leading to transfusion of two or more units of whole blood or red blood cells.
Ischemic or hemorrhagic stroke | Within 7 days and 30 days
All-cause mortality | Within 7 days, 30 days, 6 months, and 12 months
  Death due to any cause
Serious adverse events | Within 30 days
All-cause mortality, cardiorespiratory collapse or recurrence of PE | Within 30 days
  Death due to any cause,
  Cardiorespiratory collapse or decompensation should fulfill at least one of the following criteria:
  1. cardiac arrest or need for CPR at any time between randomization and day 7;
  2. signs of shock: new-onset persistent arterial hypotension (SBP below 90 mmHg or SBP drop by at least 40 mmHg over at least 15 minutes, and despite an adequate filling status; or need for vasopressors to maintain SBP of at least 90 mmHg), accompanied by end-organ hypoperfusion (altered mental status; oliguria/anuria; or increased serum lactate) at any time between randomization and day 7;
  3. placement on ECMO at any time between randomization and day 7;
  4. intubation, or initiation of non-invasive mechanical ventilation at any time between randomization and day 7;
  5. National Early Warning Score (NEWS) of 9 or higher, between 24 hours and 7 days after randomization, confirmed on consecutive measurements, taken twice.
Symptomatic PE recurrence | Within 30 days and 6 months
Change from baseline in RV dysfunction on echocardiography | 6 months
  Right ventricle to left ventricle end diastolic diameter ratio (RV/LV)
Duration of hospitalization for the index PE event | Within 30 days
  Time from admission to discharge from hospital
Duration of stay at the intensive, intermediate or coronary care unit during hospitalization for the index PE event | Within 30 days
  Time from admission to discharge from ICU, intermediate, or ICC
Functional status as measured by World Health Organization (WHO) functional class | Up to 7 days, 30 days, 6 and 12 months
  The World Health Organization (WHO) Functional Class assessment is a system for assessing the severity of dyspnea in patients with pulmonary hypertension. Subjects will be classified as Class 1-4 at time points throughout their participation in the study.
Functional status as measured by 6-Minute Walk Test (6MWT) | 30 days, 6 and 12 months
  The 6MWT measures the distance a patient can walk on a flat surface in a period of 6 minutes. A 100 meter distance is measured in a hallway and the patient is asked to walk quickly as many laps as they can over the course of the timed test. The total distance is measured. The patient's baseline vitals and symptoms are compared to their condition at the completion of the test.
Functional status as measured by Post-Venous Thromboembolism Functional Status (PVFS) scale | 30 days, 6 and 12 months
  The Post-Venous Thromboembolism (VTE) Functional Status (PVFS) scale focuses on relevant aspects of daily life during follow-up after a venous thromboembolic event. The scale is neither intended to solely focus on VTE-associated functional limitations nor to diagnose post-VTE syndrome. In contrast, the scale has been developed to help users become aware of current functional limitations in patients who have suffered a VTE, whether or not as a result of the specific VTE, and to objectively determine the degree of disability,
Quality of life using PEmb-QOL | 6 and 12 months
  PEmb-QOL is a questionnaire that assesses post-pulmonary embolism quality of life in the context of pulmonary-specific symptoms. The PEmb-QOL questionnaire contains six dimensions based on the contents of the items: frequency of complaints, limitations in activities of daily living, work-related problems, social limitations, intensity of complaints and emotional complaints. Higher scores indicate worse outcome.
Quality of life using SF-36 | 6 and 12 months
  The SF-36 questionnaire is a generic quality of life measure containing eight health domains (physical functioning, physical role, pain, general health, vitality, social function, emotional role functioning, and mental health). The scoring is on a 0-100 scale, with a higher score indicating better health. Scores are combined into two overall summary scores: physical health summary score and mental health summary score.
Quality of life using EQ-5D scale | 6 and 12 months
  The EQ-5D is a patient reported outcome that provides a simple descriptive profile and single index value for health status. The questionnaire consists of 5 questions pertaining to specific health dimensions, including mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and overall health status rating scale.
Diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH) | Within 12 months
  CTEPH will be diagnosed by the investigational site according to presence of all of the following criteria:
  1. At least one mismatched segmental perfusion defect demonstrated by ventilation/perfusion scanning after 3 months of adequate therapeutic anticoagulation
  2. Resting mean pulmonary arterial pressure (mPAP) ≥25 mmHg measured by invasive right heart catheterization
  3. Pulmonary capillary wedge pressure ≤15 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Konstantinides, MD, Principal Investigator — University Medical Center Mainz, Mainz, Germany; Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital, Boston, Massachusetts, USA
Locations (62):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Christiana Hospital, Newark, Delaware
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Methodist Hospitals, Merrillville, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health East Louisville, Lousville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital - University Medical Center, Camden, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Kettering Health, Kettering, Ohio
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Medical Center, Austin, Texas
  - Houston Methodist Sugarland Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Wisconsin Hospitals, Madison, Wisconsin
- Austria (4):
  - A.o. LKH Univ.-Kliniken Innsbruck, Innsbruck
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Allgemeines Krankenhaus AKH, Vienna
  - Austria Klinik Ottakring Vienna, Vienna
- France (3):
  - CHU de Besancon, Besançon
  - CHU (Nimes Cedex), Nîmes
  - Hôpital Européen Georges Pompidou (HEGP), Paris
- Germany (11):
  - Uniklinik Aachen, Aachen
  - Klinikum Bielefeld, Bielefeld
  - GFO Kliniken Bonn, Bonn
  - Klinikum Chemnitz, Chemnitz
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinik Immenstadt, Immenstädt
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Klinikum Rechts der Isar, Munich
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Galway, Galway
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Universitair Medisch Centrum, Utrecht
- Poland (3):
  - John Paul II Hospital, Krakow
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Medical University of Warsaw, Warsaw
- Switzerland (3):
  - University Hospital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - The Royal Free Hospital, London
  - Northwick Park Hospital, Middlesex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barco S, Vicaut E, Klok FA, Lankeit M, Meyer G, Konstantinides SV; PEITHO Investigators. Improved identification of thrombolysis candidates amongst intermediate-risk pulmonary embolism patients: implications for future trials. Eur Respir J. 2018 Jan 18;51(1):1701775. doi: 10.1183/13993003.01775-2017. Print 2018 Jan. No abstract available. PMID 29348184
- [Background] Marti C, John G, Konstantinides S, Combescure C, Sanchez O, Lankeit M, Meyer G, Perrier A. Systemic thrombolytic therapy for acute pulmonary embolism: a systematic review and meta-analysis. Eur Heart J. 2015 Mar 7;36(10):605-14. doi: 10.1093/eurheartj/ehu218. Epub 2014 Jun 10. PMID 24917641
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Becattini C, Agnelli G, Lankeit M, Masotti L, Pruszczyk P, Casazza F, Vanni S, Nitti C, Kamphuisen P, Vedovati MC, De Natale MG, Konstantinides S. Acute pulmonary embolism: mortality prediction by the 2014 European Society of Cardiology risk stratification model. Eur Respir J. 2016 Sep;48(3):780-6. doi: 10.1183/13993003.00024-2016. Epub 2016 May 12. PMID 27174887
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Bajaj NS, Kalra R, Arora P, Ather S, Guichard JL, Lancaster WJ, Patel N, Raman F, Arora G, Al Solaiman F, Clark DT 3rd, Dell'Italia LJ, Leesar MA, Davies JE, McGiffin DC, Ahmed MI. Catheter-directed treatment for acute pulmonary embolism: Systematic review and single-arm meta-analyses. Int J Cardiol. 2016 Dec 15;225:128-139. doi: 10.1016/j.ijcard.2016.09.036. Epub 2016 Sep 20. PMID 27718446
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Steering Committee. Single-bolus tenecteplase plus heparin compared with heparin alone for normotensive patients with acute pulmonary embolism who have evidence of right ventricular dysfunction and myocardial injury: rationale and design of the Pulmonary Embolism Thrombolysis (PEITHO) trial. Am Heart J. 2012 Jan;163(1):33-38.e1. doi: 10.1016/j.ahj.2011.10.003. PMID 22172434
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] GUSTO investigators. An international randomized trial comparing four thrombolytic strategies for acute myocardial infarction. N Engl J Med. 1993 Sep 2;329(10):673-82. doi: 10.1056/NEJM199309023291001. PMID 8204123
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Liu VX, Lu Y, Carey KA, Gilbert ER, Afshar M, Akel M, Shah NS, Dolan J, Winslow C, Kipnis P, Edelson DP, Escobar GJ, Churpek MM. Comparison of Early Warning Scoring Systems for Hospitalized Patients With and Without Infection at Risk for In-Hospital Mortality and Transfer to the Intensive Care Unit. JAMA Netw Open. 2020 May 1;3(5):e205191. doi: 10.1001/jamanetworkopen.2020.5191. PMID 32427324
- [Background] Smith GB, Prytherch DR, Meredith P, Schmidt PE, Featherstone PI. The ability of the National Early Warning Score (NEWS) to discriminate patients at risk of early cardiac arrest, unanticipated intensive care unit admission, and death. Resuscitation. 2013 Apr;84(4):465-70. doi: 10.1016/j.resuscitation.2012.12.016. Epub 2013 Jan 4. PMID 23295778
- [Background] Quiroz R, Kucher N, Schoepf UJ, Kipfmueller F, Solomon SD, Costello P, Goldhaber SZ. Right ventricular enlargement on chest computed tomography: prognostic role in acute pulmonary embolism. Circulation. 2004 May 25;109(20):2401-4. doi: 10.1161/01.CIR.0000129302.90476.BC. Epub 2004 May 17. PMID 15148278
- [Background] Stein PD, Matta F, Yaekoub AY, Goodman LR, Sostman HD, Weg JG, Hales CA, Hull RD, Leeper KV Jr, Beemath A, Saeed IM, Woodard PK. Reconstructed 4-chamber views compared with axial imaging for assessment of right ventricular enlargement on CT pulmonary angiograms. J Thromb Thrombolysis. 2009 Oct;28(3):342-7. doi: 10.1007/s11239-009-0331-5. Epub 2009 Mar 27. PMID 19326189
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Klok FA, Cohn DM, Middeldorp S, Scharloo M, Buller HR, van Kralingen KW, Kaptein AA, Huisman MV. Quality of life after pulmonary embolism: validation of the PEmb-QoL Questionnaire. J Thromb Haemost. 2010 Mar;8(3):523-32. doi: 10.1111/j.1538-7836.2009.03726.x. Epub 2009 Dec 15. PMID 20025645
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Burnett AE, Mahan CE, Vazquez SR, Oertel LB, Garcia DA, Ansell J. Guidance for the practical management of the direct oral anticoagulants (DOACs) in VTE treatment. J Thromb Thrombolysis. 2016 Jan;41(1):206-32. doi: 10.1007/s11239-015-1310-7. PMID 26780747
- [Background] Cech DJ, Martin ST. Evaluation of function, activity, and participation. Functional Movement Development Across the Life Span (Third Edition), 2012.
- [Background] Saris-Baglama RN, Dewey CJ, Chisholm GB, et al. QualityMetric health outcomes™ scoring software 4.0. Lincoln, RI: QualityMetric Incorporated, 2010, p. 138.
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Derived] Klok FA, Piazza G, Sharp ASP, Ni Ainle F, Jaff MR, Chauhan N, Patel B, Barco S, Goldhaber SZ, Kucher N, Lang IM, Schmidtmann I, Sterling KM, Becker D, Martin N, Rosenfield K, Konstantinides SV. Ultrasound-facilitated, catheter-directed thrombolysis vs anticoagulation alone for acute intermediate-high-risk pulmonary embolism: Rationale and design of the HI-PEITHO study. Am Heart J. 2022 Sep;251:43-53. doi: 10.1016/j.ahj.2022.05.011. Epub 2022 May 16. PMID 35588898